CLINICAL TRIAL: NCT04312958
Title: Evaluation of the Clinical Performance of the Quantra System With the QStat Cartridge in Trauma and Liver Transplantation
Brief Title: Quantra QStat in Trauma and Liver Transplant
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-032
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hemorrhage; Trauma; Liver Transplant
Keywords: Viscoelastic testing; Coagulation; Trauma; Liver Transplant; Quantra; QStat
MeSH Terms: conditions — Hemorrhage; Wounds and Injuries; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Trauma patients: Trauma patients experiencing traumatic injuries requiring a full trauma team response.
  Interventions: Diagnostic Test: Quantra System
- Liver transplant patients: Patients undergoing liver transplant surgery.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care.
  Other Names: Quantra QStat Cartridge

SUMMARY:
This is a multi-center prospective, observational study of the Quantra System with the QStat Cartridge in trauma patients and patients undergoing liver transplant.

DETAILED DESCRIPTION:
The Quantra System is a fully integrated and automated in vitro diagnostic device which uses SEER Sonorheometry, an ultrasound-based technology, to characterize the viscoelastic properties of a whole blood sample during coagulation. The QStat Cartridge was developed to monitor hemostasis in patients that may experience a range of coagulopathies of various etiologies, including fibrinolytic defects. These patients include the trauma and liver transplant populations. The cartridge consists of four independent channels each containing different sets of reagents, which provide four measurements performed in parallel yielding five parameters that depict the functional status of a patient's coagulation system.

This multi-center, prospective, observational pilot study will evaluate the performance of the Quantra System with the QStat Cartridge as compared to conventional viscoelastic testing methods in blood samples obtained from trauma patients and patients undergoing liver transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years
* Subject is a trauma patient experiencing traumatic injuries requiring a full trauma team response OR Subject is a patient undergoing liver transplant surgery.
* Subject, or subject's legally authorized representative (LAR), is willing to provide informed consent, either prospectively or by deferred consent, OR Institutional Review Board (IRB)/Ethics Committee (EC) has waived the requirement to obtain informed consent.

Exclusion Criteria:

* Subject is younger than 18 years of age
* Subject is pregnant.
* Subject is incarcerated at the time of the study.
* Subject is currently enrolled in a distinct study that might confound the result of the proposed study
* Subject is affected by a condition that, in the opinion of the surgical team, may pose additional risks.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Potential study participants will be adult (>18 years) trauma patients or patients undergoing liver transplant surgery.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Comparison of Quantra Clot Time (CT) to ROTEM Delta INTEM CT results | Upon arrival of trauma subject to the emergency department
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Time (CT) to ROTEM Delta INTEM CT results | Baseline, immediately before the start of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Time (CT) to ROTEM Delta INTEM CT results | During anhepatic phase of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Time (CT) to ROTEM Delta INTEM CT results | During post-reperfusion phase of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Stiffness (CS) to ROTEM Delta EXTEM A20 results | Upon arrival of trauma subject to the emergency department
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Stiffness (CS) to ROTEM Delta EXTEM A20 results | Baseline, immediately before the start of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Stiffness (CS) to ROTEM Delta EXTEM A20 results | During anhepatic phase of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Stiffness (CS) to ROTEM Delta EXTEM A20 results | During post-reperfusion phase of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Fibrinogen Contribution (FCS) to ROTEM Delta FIBTEM A20 results | Upon arrival of trauma subject to the emergency department
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Fibrinogen Contribution (FCS) to ROTEM Delta FIBTEM A20 results | Baseline, immediately before the start of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Fibrinogen Contribution (FCS) to ROTEM Delta FIBTEM A20 results | During anhepatic phase of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Fibrinogen Contribution (FCS) to ROTEM Delta FIBTEM A20 results | During post-reperfusion phase of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Stability to Lysis (CSL) to ROTEM Delta EXTEM ML results | Upon arrival of trauma subject to the emergency department
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Stability to Lysis (CSL) to ROTEM Delta EXTEM ML results | Baseline, immediately before the start of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Stability to Lysis (CSL) to ROTEM Delta EXTEM ML results | During anhepatic phase of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta
Comparison of Quantra Clot Stability to Lysis (CSL) to ROTEM Delta EXTEM ML results | During post-reperfusion phase of liver transplant surgery
  Coagulation function assessed by Quantra and ROTEM Delta

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - University of Colorado, Denver, Colorado
  - University of Florida Health Shands Hospital, Gainesville, Florida
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Ohio State University, Columbus, Ohio
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moore EE, Michelson EA, Gabriel-Ramos K, Cripps MW, Flores A, Vandyck K, Thurston B, Brennan M, Viola F, Winegar DA. Multicenter evaluation of the Quantra with the QStat Cartridge in adult trauma patients. Trauma Surg Acute Care Open. 2025 Jun 3;10(2):e001672. doi: 10.1136/tsaco-2024-001672. eCollection 2025. PMID 40486089